CLINICAL TRIAL: NCT07005323
Title: Phase I/IIa Clinical Study of PAL-222 Targeting Patients With Neovascular Age-related Macular Degeneration (AMD) That Shows no Response to Existing Therapy
Brief Title: Progression Suppression and Retinal Regression in VEGF-resistant AMD
Acronym: PRESERVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: PharmaBio Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAL-222-P2
Record Dates: First submitted 2025-03-03; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Neovascular Age-related Macular Degeneration (AMD)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Therapeuitic group (Experimental): One sheet of PAL-222 is implanted into the subretinal space of either of eyes through pars plana vitrectomy.
  Interventions: Procedure: Pars plana vitrectomy

INTERVENTIONS:
Procedure: Pars plana vitrectomy — One sheet of PAL-222 is implanted into the subretinal space of either of eyes through pars plana vitrectomy.

SUMMARY:
The goal of this clinical trial is to assess safety and efficacy in patients with Neovascular Age-related Macular Degeneration with no response to existing therapy.

The main measures it aims to answer are:

* Investigation of adverse events
* Changes in clinical testing data
* Changes in vital signs
* Changes in intraocular pressure of the therapeutic eye
* Changes in testing of anterior segment of the therapeutic eye Participants will be implanted one sheet of PAL-222 into the subretinal space through pars plana vitrectomy.

Researchers will compare pre and post implantation of therapeutic eye to see if any safety issues recognized

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 50 and 85 years at the time of consent acquisition
2. Patients diagnosed neovascular AMD in one or both eyes
3. Patients with corrected letter vision in the subject eye of 20 letters or more (equivalent to decimal vision of 0.05) and less than 60 letters (equivalent to decimal vision of 0.32)
4. Patients who apply to one or more of the followings:

   ① RPE defect site in the RPE tear includes the Fovea

   ② The Macular atrophy confirmed by low fundus autofluorescence extends to the fovea

   ③ Patients with choroidal thinning (150 micrometer and less), subretinal fluid resistant to standard treatment, and high activity, but without hard exudated or subretinal hemorrhage which are indicators of the high risk of visual impairment.

   ④ Patients with cystoid macular degeneration with photoreceptor cell loss and intraretinal fluid above fibrovascular pigment epithelial detachment, but without hard exudates or subretinal hemorrhage.
5. Patients who had little improvement in exudative changes and no improvement, or deterioration of vision in recent two treatment with VEGF inhibitor therapy (two consecutive administration at 4-8-week intervals), after existing therapy

Exclusion Criteria:

1. Patients with fibrovascular pigment epithelial detachment (thickness 50 µm or more) in the subfoveal area in the subject eye.
2. Patients with hard exudates in the subretinal or intraretinal area in the subject eye.
3. Patients with eye infections
4. Patients with a history of retinal vascular disease other than neovascular AMD, retinal degenerative disease, rhegmatogenous retinal detachment, macular hole, premacular membrane with retinal wall, uveitis, or other ocular inflammatory disease in the subject eye.
5. Patients with optic nerve atrophy in the subject eye
6. Patients with progressive glaucoma in the subject eye (in whom intraocular pressure is not controlled, or visual field loss is progressive or has already spread to the macula)
7. Patients with severe myopia in the subject eye (axial length of 26.5 mm or more, or spherical equivalent of -7.0 D or less in phakic eyes)
8. Patients who have undergone intraocular surgery in the subject eye. (In the case of cataract surgery, patients may be enrolled if they have had no endophthalmitis or other complications, have progressed well, and more than 3 months have passed since the surgery)
9. Patients with corrected visual acuity of the non-subject eye 0.1 or less
10. Patients who are currently receiving or will receive VEGF inhibitor treatment in the non-subject eye during the study period
11. Patients with abnormal findings that pose a problem in clinical trial participation in screening tests.
12. Patients with positive HBs antigen, HCV antibody, HIV antibody, HTLV-1 antibody, syphilis serum reaction
13. Patients with allergies to human serum albumin antibiotics, trypsin
14. Patients with severe blood disorders, heart failure, liver disorders, and renal disorders
15. Patients diagnosed with malignant tumor within 5 years or patients requiring treatment
16. Pregnant women, lactating women, patients wishing to become pregnant during the trial period
17. Patients who cannot discontinue anticoagulants or antiplatelet drugs before the trial
18. Patients with drug addiction or alcoholism

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Safety Evaluation: Incidence, type, and severity of Adverse Events (AE) | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hitoshi Kusano, M.D., Study Chair — PhamaBio Coorporation
Locations (1):
- Yamaguchi University Hospital, Ube, Ymaguchi, Japan

IPD SHARING:
Plan to Share IPD: No